CLINICAL TRIAL: NCT01346995
Title: The Effect of Experimental Knee Pain During Strengthening Exercises on Muscle Strength Gain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Frederiksberg University Hospital (Other)
Responsible Party: Henning Bliddal, The Parker Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 072.07
Record Dates: First submitted 2011-05-02; First posted 2011-05-04 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2010-02

CONDITIONS: Muscle Strength

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Knee Pain (Experimental): Experimental knee pain induced by injections of 1 ml hypertonic saline in to the infrapatellar fat pad
  Interventions: Other: Experimental knee pain
- Control (Active Comparator): non-painful injections of isotonic saline into the infrapatellar fatpad.
  Interventions: Other: Non-painful control injections

INTERVENTIONS:
Other: Experimental knee pain — Injection of 1 ml hypertonic saline (5.8%) into the infrapatellar fat pad
  Arms: Experimental Knee Pain
Other: Non-painful control injections — Injection of isotonic saline into the infrapatellar fat pad
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the effects of experimental knee pain on the muscle strength gain after 8 weeks of strengthening exercises for the quadriceps. It is hypothesized that experimental knee pain will reduce the muscle strength gain following strengthening exercises in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* aged between 20 to 35 years
* healthy
* untrained (non-regular exercise participation [i.e. < 1 day/week])

Exclusion Criteria:

* symptomatic musculoskeletal diseases
* history of traumatic injuries to muscles, tendons or joints of the lower extremity
* knee joint pain within a month prior to enrollment

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2010-02; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Isokinetic knee muscle strength | At baseline and after 8 weeks of exercise

SECONDARY OUTCOMES:
One-leg chair rise | At baseline and after 8 weeks of exercise

REFERENCES:
- [Derived] Sorensen TJ, Langberg H, Hodges PW, Bliddal H, Henriksen M. Experimental knee joint pain during strength training and muscle strength gain in healthy subjects: a randomized controlled trial. Arthritis Care Res (Hoboken). 2012 Jan;64(1):108-16. doi: 10.1002/acr.20618. PMID 21905254